CLINICAL TRIAL: NCT04144491
Title: A Nutritional Trial on Effect of Probiotic Yoghurt Containing Lactobacillus Rhamnosus Yoba on Respiratory Tract Infection and Other Health Outcomes Among Children Aged 3-6 Years in Southwest Uganda
Brief Title: Effect of L. Rhamnosus Yoba on RTI and Other Health Outcomes Among Children (3-6 Years) in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Collaborators: Yoba for Life Foundation (Unknown)
Responsible Party: Principal Investigator, Remco Kort, Professor, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 01/09-19
Record Dates: First submitted 2019-09-14; First posted 2019-10-30 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Respiratory Tract Infections; Diarrhea; Skin Diseases; Tinea Capitis; Common Cold
Keywords: Lactobacillus rhamnosus yoba 2012; Children
MeSH Terms: conditions — Respiratory Tract Infections; Diarrhea; Skin Diseases; Tinea Capitis; Common Cold | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoghurt (Experimental): Yoghurt, containing Lactobacillus rhamnosus yoba 2012, Streptococcus thermophilus C104, whole milk, 5% sugar, 0.1% strawberry or vanilla flavor essence.
  Interventions: Dietary Supplement: Probiotic
- Custard (Placebo Comparator): Custard, containing whole milk, 5% sugar, 0.1% strawberry or vanilla flavor essence, 4% modified corn starch.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotics are defined by the Food and Agricultural Organization (FAO)/WHO as "live microorganisms, which when consumed in adequate amounts, confer a health benefit on the host". Lactobacillus rhamnosus GG (LGG) is the most documented probiotic bacteria, with many proven unique characteristics and therewith associated health benefits. No adverse effects of the consumption of LGG in healthy infants have been reported. The Lactobacillus rhamnosus yoba containing yoghurt drink, which is locally produced and subsequently consumed by resource-poor communities in rural Uganda has been described. The strain used in this intervention is a generic variant of LGG, called Lactobacillus rhamnosus yoba 2012. LGG is consumed as part of food all over the world, and is not a drug.
  100ml of yoghurt containing Lactobacillus rhamnosus yoba 2012 will be consumed 5 days per week, for 9 weeks.
  Other Names: Lactobacillus rhamnosus yoba 2012; Lactobacillus rhamnosus GG
  Arms: Yoghurt
Dietary Supplement: Placebo — 100ml of custard will be consumed 5 days per week, for 9 weeks.
  Arms: Custard

SUMMARY:
This is a nutritional trial with two arms: 1) Intervention arm of Probiotic Yoghurt containing Lactobacillus rhamnosus yoba 2012 and 2) Control arm of custard-like dairy product. The study subjects are 200 children between the age of 3-6 years that attend a school in Southwestern Uganda, Sheema district. Children will be randomized and enrolled in either the yoghurt (100 children) or the placebo (100 children) arm. The children will be monitored for 3 weeks in the baseline in regards to the incidence of common childhood diseases. During these three weeks, stool, saliva and urine samples will be collected. Also measurement of anthropometric indicators (weight and height) will take place. Subsequently, the children will consume either 100ml yoghurt or 100ml placebo product, once per day for five days per week for nine weeks, while being daily monitored in regards to the incidence of common childhood diseases. The same samples (stool, urine and saliva) and assessments (anthropometric) will take place at end line.

DETAILED DESCRIPTION:
This is a nutritional trial with two arms: 1) Intervention arm of Probiotic Yoghurt containing Lactobacillus rhamnosus yoba 2012 and 2) Placebo arm of custard-like dairy product. The study subjects are 200 children between the age of 3-6 years that attend a school in Southwestern Uganda, Sheema district. Children will be randomized and enrolled in either the yoghurt (100 children) or the placebo (100 children) arm. The children will be monitored for 3 weeks in the baseline in regards to the incidence of common childhood diseases. During these three weeks, stool, saliva and urine samples will be collected. Also measurement of anthropometric indicators (weight and height) will take place. Subsequently, the children will consume either 100ml yoghurt or 100ml placebo product, once per day for five days per week for nine weeks, while being daily monitored in regards to the incidence of common childhood diseases. The same samples (stool, urine and saliva) and assessments (anthropometric) will take place at end line. The yoghurt and the placebo product will be locally sourced in the district where the school is located. Monitoring and data collection tools are:

1. Baseline, mid line and end line questionnaire administered to parents to identify confounding factors (e.g. use of medication and diet from home) of treatment and control group.
2. Weight and height measurements at baseline and end line in both the treatment and control group (total 2 times).
3. Daily monitoring of the incidence of RTIs, diarrhoea, skin rashes or other diseases in treatment and control groups by a nurse, registered in a mobile application.
4. Collection of urine samples every 4 weeks for 3 months (total 4 times), for assessment of impact of the intervention on system health.
5. Collection of stool samples at baseline and end line, for assessment of impact of the intervention on gut health.
6. Collection of saliva samples before and towards the end of the intervention, for assessment of impact of the intervention on immune biomarkers

The consumption of probiotic yoghurt at school as paid for by the parents, is currently being promoted by an Non-Governmental Organization (NGO) in the region. Following this program, children from a primary school that includes a pre-primary section, in which both the management and the parents have recently decided to purchase yoghurt for the pupils on regular basis will be recruited. The study subjects (children) are recruited at these institutions, after consent from the parent has been obtained. The parent is free to provide his/her child with yoghurt, even if the parent does not consent for the child to take part in the study.

The study will start three weeks before either yoghurt or placebo consumption commences, in order to establish a solid baseline. With the help of tablets and a specially designed mobile application, nurses will keep track of their pupils' health by tracking incidence of diarrhoea, respiratory tract infections, skin rashes and other diseases. Teachers will keep track of the daily attendance of pupils.

Measurements of weight and height will be measured by a nurse at baseline and end line. The measurements will be conducted with the help of Standard Operations Procedures as provided by Life Study and analyzed with the help of World Health Organization (WHO) guidelines. Urine samples will be taken from the children at baseline, after 4 weeks, after 8 weeks, and at end line (12 weeks). Stool samples and saliva samples will be taken at the beginning and the end of the study.

During these 3 months in which the children will be monitored, a questionnaire will be administered to the parents of the children at the start, middle and end of the study. The primary objective and content of the questionnaire is related to diet of the children outside school, in order to determine whether there are significant differences between the diets of the children in the treatment group and in the control group. The questionnaires will furthermore include questions about absenteeism and causes thereof, incidence of diarrhoea, Respiratory Tract Infections (RTI) or any other diseases, and the use of any type of drug or treatment, in order to verify and supplement the information provided by the class-teacher. Lastly, information on the vaccination history of the child will be obtained from the parent

ELIGIBILITY:
Inclusion Criteria:

* Children of a pre-primary institution in Southwest Uganda are targetted
* During interactions with the pre-primary institutions prior to the study, the parents of the children have agreed to pay for their child to either take probiotic yoghurt (100ml five times per week).
* Parents are willing to provide written consent for their child to participate in the study

Exclusion Criteria:

* The child does not comply with the inclusion criteria
* The child has an aversion against yoghurt or milk products
* The child is lactose-intolerant as indicated by the parent, or has any other medical condition that will prevent him/her from taking yoghurt or milk products

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 195 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
The number of children on each individual day that suffers from Respiratory Tract Infections | 3 months
  To compare the incidence of respiratory tract infections among children aged 3-6 years in Southwest Uganda before, during and after an intervention with probiotic yoghurt containing Lactobacillus rhamnosus yoba

SECONDARY OUTCOMES:
Changes in weight of children during the study period | 3 months
  To monitor changes in weight of children aged 3-6 years in Southwest Uganda who consume yoghurt containing Lactobacillus rhamnosus yoba.
Changes in height of the children during the study period | 3 months
  To monitor changes in height of children aged 3-6 years in Southwest Uganda who consume yoghurt containing Lactobacillus rhamnosus yoba.
The number of children on each individual day that suffers from Diarrhea | 3 months
  To compare the incidence of diarrhea among the children before, during and after the intervention.
The number of children on each individual day that suffers from any form of skin diseases | 3 months
  To compare the incidence of skin rashes among the children before, during and after the intervention.
The number of children on each individual day that is absent | 3 months
  To compare absenteeism as a result of sickness among the children before, during and after the intervention.
Differences in the metabolic profile of childrens urine between baseline and after 9 weeks of intervention using 1H-Nuclear Magnetic Resonance (NMR) Spectroscopy | 3 months
  To compare metabolic profile in the urine of the children before, during and after the intervention
Differences in the microbial profile of childrens stool between baseline and after 9 weeks of intervention using Next Generation Sequencing (NGS) in combination with Fluorescence In Situ Hybridisation hyphenated to Flow Cytometry (Flow-FISH) | 3 months
  To compare the microbial profile in the stool of the children before and after the intervention.
Differences in the immune markers of childrens saliva between baseline and after 9 weeks of intervention | 3 months
  To compare immune markers (secretory immunoglobulin A (IgA), secretory leukoprotease inhibitor (SLPI), immunoglobulin M (IgM), immunoglobulin G (IgG), cytokines chemokines and growth factors) in the saliva of the children before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Remco Kort, PhD, Principal Investigator — VU Amsterdam
Locations (1):
- Paragon primary and nursery School, Kabwohe, Sheema, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dezateux, C., Williams, J., Walton, S., Wells, J., 2016. Life Study Standard Operating Procedures: Adult Anthropometry.
- [Background] Williams, J., Walton, S., Wells, J., 2016. Life Study Standard Operating Procedures: Infant Anthropometry.
- [Background] World Health Organization (Ed.), 2007. WHO child growth standards: head circumference-for-age, arm circumference-for-age, triceps skinfold-for-age and subscapular skinfold-for-age: methods and development. World Health Organization, Geneva
- [Background] World Health Organization (Ed.), 2006. WHO child growth standards: length/height-for-age, weight-for-age, weight-for-length, weight-for-height and body mass index-for-age ; methods and development. WHO Press, Geneva.
- [Background] Pineiro M, Stanton C. Probiotic bacteria: legislative framework-- requirements to evidence basis. J Nutr. 2007 Mar;137(3 Suppl 2):850S-3S. doi: 10.1093/jn/137.3.850S. PMID 17311986
- [Background] Petschow BW, Figueroa R, Harris CL, Beck LB, Ziegler E, Goldin B. Effects of feeding an infant formula containing Lactobacillus GG on the colonization of the intestine: a dose-response study in healthy infants. J Clin Gastroenterol. 2005 Oct;39(9):786-90. doi: 10.1097/01.mcg.0000177245.53753.86. PMID 16145341
- [Background] Scalabrin D, Harris C, Johnston WH, Berseth CL. Long-term safety assessment in children who received hydrolyzed protein formulas with Lactobacillus rhamnosus GG: a 5-year follow-up. Eur J Pediatr. 2017 Feb;176(2):217-224. doi: 10.1007/s00431-016-2825-4. Epub 2016 Dec 15. PMID 27975116
- [Background] Kort R, Westerik N, Mariela Serrano L, Douillard FP, Gottstein W, Mukisa IM, Tuijn CJ, Basten L, Hafkamp B, Meijer WC, Teusink B, de Vos WM, Reid G, Sybesma W. A novel consortium of Lactobacillus rhamnosus and Streptococcus thermophilus for increased access to functional fermented foods. Microb Cell Fact. 2015 Dec 8;14:195. doi: 10.1186/s12934-015-0370-x. PMID 26643044
- [Background] Kort R, Sybesma W. Probiotics for every body. Trends Biotechnol. 2012 Dec;30(12):613-5. doi: 10.1016/j.tibtech.2012.09.002. Epub 2012 Sep 29. No abstract available. PMID 23031355